CLINICAL TRIAL: NCT00700427
Title: Maintenance of Response After Open-Label Treatment With Atomoxetine Hydrochloride in Adult Outpatients With Attention-Deficit/Hyperactivity Disorder (ADHD): A Placebo-Controlled, Randomized Withdrawal Study
Brief Title: A Long Term Study of a Medication for Adults With Attention-Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9655; B4Z-MC-LYDO (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-06-16; First posted 2008-06-18 (Estimated); Results first posted 2013-05-29 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Adult; long term; maintenance of response; Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atomoxetine (Experimental): Atomoxetine 40-100 milligrams per day (mg/day) orally, once daily or twice daily for 24 weeks, followed by atomoxetine 80-100 mg/day orally, once daily or twice daily for 25 weeks.
  Interventions: Drug: atomoxetine hydrochloride
- Placebo (Placebo Comparator): Atomoxetine 40-100 mg/day orally, once daily or twice daily for 24 weeks, followed by placebo orally, once daily for 25 weeks.
  Interventions: Drug: atomoxetine hydrochloride; Drug: Placebo

INTERVENTIONS:
Drug: atomoxetine hydrochloride — Oral 40-100 mg/day
  Other Names: Strattera; LY139603; atomoxetine
Drug: Placebo — Oral delivery of matching placebo
  Arms: Placebo

SUMMARY:
LYDO is a multi-center study that will enroll approximately 1925 adult outpatients with Attention Deficit/Hyperactivity Disorder (ADHD). Patients will receive, under open label conditions, atomoxetine up to 100 mg/day during the acute, open-label part of the study. Those patients that meet the response criteria will continue the blind phase of the study up to a year. During that period, patients that respond to atomoxetine will be randomized to continue the treatment with atomoxetine or with placebo (neither the patients nor investigators know if patients receive atomoxetine or placebo).

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Male or female
* Must meet Attention-Deficit/Hyperactivity Disorder (ADHD) according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition Text Revision™ (DSM-IV-TR™) criteria

Exclusion Criteria:

* Comorbidity with major psychiatric disorder
* Clinically significant depression or anxiety
* Patients with significant medical conditions
* Current alcohol/drugs abuse/dependence
* Concomitant excluded medications

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2017 (Actual)
Dates: Start 2008-06; Primary Completion 2011-08 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 am - 5 pm Eastern Time (UTC/GMT - 5hours, EST), Study Director — Eli Lilly and Company
Locations (56):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna, Austria
- Belgium (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bruges
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kortenberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liège
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mechelen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Uccle
- Finland (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Helsinki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampere
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Turku
- France (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bordeaux
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Douai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marseille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montpellier
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orvault
- Germany (18):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ahrensburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bochum
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ellwangen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Essen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Freiburg im Breisgau
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fulda
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hadamar
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hagen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hanover
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Homburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leipzig
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ludwigshafen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mainz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mannheim
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Munich
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Würzburg
- Italy (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coppito
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Donà di Piave
- Netherlands (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amersfoort
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Flushing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hengelo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nijmegen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tilburg
- Portugal (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cascais
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coimbra
- Spain (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alcorcón
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pamplona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zamora
- Sweden (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Luleå
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lund
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Malmo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vaxjo
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lausanne, Switzerland
- United Kingdom (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brighton, East Sussex
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Storrington, West Sussex
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London

REFERENCES:
- [Derived] Tanaka Y, Escobar R, Upadhyaya HP. Assessment of effects of atomoxetine in adult patients with ADHD: consistency among three geographic regions in a response maintenance study. Atten Defic Hyperact Disord. 2017 Jun;9(2):113-120. doi: 10.1007/s12402-016-0212-7. Epub 2017 Jan 6. PMID 28058589
- [Derived] Upadhyaya H, Tanaka Y, Lipsius S, Kryzhanovskaya LA, Lane JR, Escobar R, Trzepacz PT, Allen AJ. Time-to-onset and -resolution of adverse events before/after atomoxetine discontinuation in adult patients with ADHD. Postgrad Med. 2015;127(7):677-85. doi: 10.1080/00325481.2015.1083394. Epub 2015 Sep 2. PMID 26329980
- [Derived] Upadhyaya H, Adler LA, Casas M, Kutzelnigg A, Williams D, Tanaka Y, Arsenault J, Escobar R, Allen AJ. Baseline characteristics of European and non-European adult patients with attention deficit hyperactivity disorder participating in a placebo-controlled, randomized treatment study with atomoxetine. Child Adolesc Psychiatry Ment Health. 2013 May 6;7(1):14. doi: 10.1186/1753-2000-7-14. PMID 23648011
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of 4 treatment periods: 12 weeks open-label, acute-treatment (trx) phase (Study Period 2), 12 weeks double-blind maintenance phase of Study Period 3 (Study Period 3A), 25 weeks double-blind randomized withdrawal phase of Study Period 3 (Study Period 3B) and an Open-Label Extension Period (Study Period 4) lasting up to 2.3 years.
Groups:
- Atomoxetine (Study Period 2): 40-100 milligrams/day (mg/day) atomoxetine orally, once daily or twice daily for 12 weeks during open-label, acute-treatment phase (Study Period 2).
- Atomoxetine (Study Period 3A): 40-100 milligrams/day (mg/day) atomoxetine orally, once daily or twice daily for 12 weeks during double-blind randomized withdrawal phase (Study Period 3).
- Atomoxetine (Study Period 3B): 80-100 mg/day atomoxetine orally, once daily or twice daily for 25 weeks during double-blind randomized withdrawal phase of Study Period 3 (Study Period 3B).
- Placebo (Study Period 3B): Placebo orally, once daily or twice daily for 25 weeks during double-blind randomized withdrawal phase of Study Period 3 (Study Period 3B).
- Atomoxetine (Study Period 4): Participants who received either atomoxetine or placebo and completed the last visit of Study Period 3 who were in countries where the adult ADHD indication for atomoxetine was not approved were allowed to participant in Study Period 4 (Open-label Extension). Participants received 40 mg/day atomoxetine orally for at least 7 days after which it was increased to 80-100 mg/day atomoxetine orally for up to 2.3 years.
Period: Study Period 2 (Open-Label Acute Trx)
Arm/Group | Atomoxetine (Study Period 2) | Atomoxetine (Study Period 3A) | Atomoxetine (Study Period 3B) | Placebo (Study Period 3B) | Atomoxetine (Study Period 4)
Started | 2017 | 0 | 0 | 0 | 0
Received at Least One Dose of Study Drug | 2011 | 0 | 0 | 0 | 0
Completed | 1006 (One participant was mistakenly recorded as completed. The reason for discontinuation is unknown.) | 0 | 0 | 0 | 0
Not Completed | 1011 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 298 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 173 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 164 | 0 | 0 | 0 | 0
Not completed — Protocol Interim Criteria Not Met | 161 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 108 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 90 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 8 | 0 | 0 | 0 | 0
Not completed — Clinical Relapse | 7 | 0 | 0 | 0 | 0
Not completed — Entry Criteria Not Met | 2 | 0 | 0 | 0 | 0
Period: Study Period 3A (Blinded Maintenance)
Arm/Group | Atomoxetine (Study Period 2) | Atomoxetine (Study Period 3A) | Atomoxetine (Study Period 3B) | Placebo (Study Period 3B) | Atomoxetine (Study Period 4)
Started | 0 | 1005 | 0 | 0 | 0
Completed | 0 | 524 | 0 | 0 | 0
Not Completed | 0 | 481 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 50 | 0 | 0 | 0
Not completed — Protocol Interim Criteria Not Met | 0 | 162 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 81 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 56 | 0 | 0 | 0
Not completed — Clinical Relapse | 0 | 49 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 41 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 32 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 3 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 0 | 0 | 0
Not completed — Missing - Not Otherwise Defined | 0 | 5 | 0 | 0 | 0
Period: Study Period 3B (Randomized Withdrawal)
Arm/Group | Atomoxetine (Study Period 2) | Atomoxetine (Study Period 3A) | Atomoxetine (Study Period 3B) | Placebo (Study Period 3B) | Atomoxetine (Study Period 4)
Started | 0 | 0 | 266 | 258 | 0
Completed | 0 | 0 | 184 | 165 | 0
Not Completed | 0 | 0 | 82 | 93 | 0
Not completed — Adverse Event | 0 | 0 | 8 | 5 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 25 | 34 | 0
Not completed — Protocol Violation | 0 | 0 | 23 | 25 | 0
Not completed — Lost to Follow-up | 0 | 0 | 19 | 9 | 0
Not completed — Lack of Efficacy | 0 | 0 | 3 | 11 | 0
Not completed — Protocol Interim Criteria Not Met | 0 | 0 | 0 | 5 | 0
Not completed — Clinical Relapse | 0 | 0 | 0 | 3 | 0
Not completed — Missing | 0 | 0 | 1 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 2 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0
Period: Study Period 4 (Open-Label Extension)
Arm/Group | Atomoxetine (Study Period 2) | Atomoxetine (Study Period 3A) | Atomoxetine (Study Period 3B) | Placebo (Study Period 3B) | Atomoxetine (Study Period 4)
Started | 0 | 0 | 0 | 0 | 180
Completed | 0 | 0 | 0 | 0 | 96
Not Completed | 0 | 0 | 0 | 0 | 84
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 16
Not completed — Death | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 12
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 38
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 2
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 2
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 11
Not completed — Clinical Relapse | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Atomoxetine (40-100 mg): 40-100 milligrams/day (mg/day) atomoxetine orally, once daily or twice daily for 12 weeks during open-label, acute-treatment period (Study Period 2).
Arm/Group | Atomoxetine (40-100 mg)
Number analyzed (Participants) | 2017
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.15 (9.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 833
  Male | 1184
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 1765
  African | 56
  Hispanic | 159
  Native American | 6
  East Asian | 14
  West Asian | 15
  Missing | 2
Region of Enrollment [Number; unit: participants]
  Argentina | 27
  Austria | 109
  Belgium | 137
  Canada | 60
  Denmark | 15
  Finland | 52
  France | 65
  Germany | 434
  Italy | 32
  Mexico | 53
  Netherlands | 71
  Portugal | 3
  Puerto Rico | 52
  Russian Federation | 6
  Spain | 153
  Sweden | 112
  Switzerland | 7
  United Kingdom | 27
  United States | 602

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Maintain a Satisfactory Response During the Double-Blind Maintenance/Randomized Withdrawal Period
Description: Conners' Adult ADHD Rating Scale-Investigator Rated:Screening Version (CAARS-Inv:SV); 30-item scale (3 subscales): inattention, hyperactivity/impulsivity (9 items each), ADHD Index (12 items). Each item is scored 0 (not at all/never) to 3 (very much/very frequently). Total ADHD symptoms score (SS)=inattention+hyperactivity/impulsivity (range:0-54). Higher score=more impairment. Clinical Global Impressions-ADHD-Severity (CGI-ADHD-S) measures participant's overall severity of ADHD symptoms and scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill participants). Maintenance of response during the randomized withdrawal phase was a reduction of ≥30% in the baseline CAARS-Inv:SV Total ADHD SS and a CGI-ADHD-S score ≤3. Participants had to continuously meet the response criteria, except for 1 excursion after assessment at Week 24 through Week 37 and 1 other excursion after assessment at Week 37 through Week 49. Excursions were not permitted at 2 consecutive visits.
Time Frame: Baseline (Week 24) up to Week 49
Population: Primary outcome measure analysis was conducted using all randomized participants in the Double-Blind Maintenance/Randomized Withdrawal Period (Study Period 3B).
Measure: Number; unit: percentage of responders
Groups:
- Atomoxetine: 80-100 milligrams/day (mg/day) atomoxetine orally, once daily or twice daily for 25 weeks during double-blind randomized withdrawal phase of Study Period 3 (Study Period 3B).
- Placebo: Placebo orally, once daily or twice daily for 25 weeks during double-blind randomized withdrawal phase of Study Period 3 (Study Period 3B).
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 266 | 258
percentage of responders | 64.3 | 50.0
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.001, Fisher Exact

2. Secondary Outcome: Number of Days Until Relapse
Description: Relapse was defined as 2 consecutive visits with a CGI-ADHD-S score ≥4 points and a return to ≥80% of participant's baseline (Visit 2) CAARS-Inv:SV Total ADHD Symptom Score (SS). If the participant showed evidence of a return of symptoms at a single visit that met severity criteria described above, and because of worsening symptoms, was unwilling to remain in the study or did not return for a second visit, the participant was also considered to have relapsed.
  CAARS-Inv:SV is a 30-item scale (3 subscales): Inattention, Hyperactivity/Impulsivity (9 items each), ADHD Index (12 items). Each item is scored 0 (0=not at all/never) to 3 (very much/very frequently). Total ADHD SS=inattention+hyperactivity/impulsivity (range: 0-54). Higher score=more impairment. CGI-ADHD-S measures participant's overall severity of ADHD symptoms and scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill participants).
Time Frame: Baseline (Week 24) up to Week 49
Population: Analyses were conducted using all randomized participants in the Double-Blind Period (Study Period 3B).
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 266 | 258
days | NA (NA) — The mean and standard deviation could not be reliably estimated because of low numbers of participants who relapsed. | NA (NA) — The mean and standard deviation could not be reliably estimated because of low numbers of participants who relapsed.

3. Secondary Outcome: Change From Baseline in the Adult Attention-Deficit/Hyperactivity Disorder (ADHD) Quality of Life (AAQoL) Scale From Week 24 to Week 49
Description: The AAQoL is a self-reported, 29-item scale assessing functional impairments in adults with ADHD. Each item is rated on a 5-point Likert scale; range: 1 (Not at all/ Never) to 5 (Extremely/Very Often). 5-domains of scale include: work functioning, family relationships, social functioning, activities of daily living (driving, managing finances), and psychological adaptation (life satisfaction, self-esteem). These scores are transformed to a 0-100 point scale (1=0; 2=25; 3=50; 4=75; 5=100), and then the item scores are summed and divided by item count to generate overall scores. The overall scores have the same total range of scores of 0-100, with higher scores indicating better quality of life. Least Squares (LS) Mean values were adjusted for baseline AAQoL score and Investigator/site.
Time Frame: Baseline (Week 24), Week 49
Population: All randomized participants with a baseline and at least 1 post-baseline AAQoL score were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 198 | 180
units on a scale | 0.4 (1.12) | -4.0 (1.10)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.002, ANCOVA

4. Secondary Outcome: Change From Baseline in Conner's Adult Attention-Deficit/Hyperactivity Disorder (ADHD) Rating Scale (Observer Rated [CAARS-O:SV]) Total ADHD Symptom Score From Week 24 to Week 49
Description: The CAARS-O:SV is a 30-item observer (typically a significant other or close friend) completed scale containing 3 subscales: inattention (9 items), hyperactivity/impulsivity (9 items), and ADHD Index (12 items). Each item is scored 0-3 (0=not at all/never; 1=just a little/once in a while; 2=pretty much/often; 3=very much/very frequently). Inattention and hyperactivity subscales range from 0-27; ADHD index subscale range is 0-36 with higher scores indicating more impaired participants. Total ADHD symptoms score=sum of the inattention and hyperactivity/impulsivity subscales, ranging from 0-54, with higher scores indicating more impaired participants. Least Squares (LS) Mean values adjusted for treatment, pooled Investigator, and baseline.
Time Frame: Baseline (Week 24), Week 49
Population: Participants with a non-missing baseline and at least 1 post-baseline CAARS-O:SV result within each group, Last Observation Carried Forward (LOCF) were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 165 | 153
units on a scale
  ADHD Imputed (Attributed) Index Score (N=164, 153) | -2.60 (0.56) | -0.10 (0.57)
  Hyperactivity/Impulsivity Subscale Imputed Score | -1.90 (0.44) | -0.10 (0.44)
  Inattention Subscale Imputed Score | -1.60 (0.46) | -0.10 (0.46)
  Total ADHD Symptom Imputed Score | -3.50 (0.83) | -0.40 (0.83)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for ADHD Imputed (Attributed) Index Score
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.002, ANCOVA — P-value for Hyperactivity/Impulsivity Subscale Imputed Score
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.009, ANCOVA — P-value for Inattention Subscale Imputed Score
Statistical Analysis 4: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.003, ANCOVA — P-value for Total ADHD Symptom Imputed Score

5. Secondary Outcome: Change From Baseline in Conner's Adult ADHD Rating Scale-Self Rated (CARRS-S:SV) Total ADHD Symptom Score From Week 24 to Week 49
Description: CAARS-S:SV is a 30-item participant completed scale containing 3 subscales: inattention (9 items), hyperactivity/impulsivity (9 items), ADHD Index (12 items). 0-3 (0=not at all/never; 1=just a little/once in a while; 2=pretty much/often; 3=very much/very frequently). Inattention and hyperactivity subscales range from 0-27; ADHD index subscale range is 0-36 with higher scores indicating more impaired participants. Total ADHD symptoms score=sum of the inattention and hyperactivity/impulsivity subscales; range: 0-54 with higher scores indicating more impaired participants. Least Squares (LS) Mean values adjusted for treatment, pooled Investigator, and baseline.
Time Frame: Baseline (Week 24), Week 49
Population: Participants with a non-missing baseline and at least 1 post-baseline CAARS-S:SV result within each treatment group, Last Observation Carried Forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 193 | 178
units on a scale
  ADHD Symptom Imputed Index Score | -1.20 (0.44) | 0.90 (0.43)
  Hyperactivity-Impulsivity Subscale Imputed Score | -0.90 (0.33) | 0.50 (0.32)
  Inattention Subscale Imputed Score | -0.70 (0.38) | 1.20 (0.37)
  Total ADHD Symptom Imputed Score | -1.60 (0.65) | 1.70 (0.64)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for ADHD Imputed (Attributed) Index Score
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Hyperactivity/Impulsivity Subscale Imputed Score
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Inattention Subscale Imputed Score
Statistical Analysis 4: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Total ADHD Symptom Imputed Score

6. Secondary Outcome: Change From Baseline in the Behavior Rating Inventory of Executive Function-Adult Version: Self Report (BRIEF-A:Self Report) Global Executive Composite (GEC) Index Score From Week 24 to Week 49
Description: The BRIEF-A:Self Report is a 75-item self-reported measure captures adults' views of their own executive functions/self-regulation in their everyday environment. Items include: Inhibit, Shift, Emotional Control, Self Monitor, Initiate, Working Memory, Plan/Organize, Task Monitor, and Organization of Materials. Behavior is rated on a 3-point scale: 1 (behavior is never observed) to 3 (behavior is often observed). GEC Index Score is a subscore of the 75-item BRIEF-A score, reflects overall functioning and was calculated based on 70 items. Total scores range: 70-210. Lower scores = less perceived impairment. Least Squares (LS) Mean values were adjusted for treatment, pooled Investigator, and baseline.
Time Frame: Baseline (Week 24), Week 49
Population: Participants with a non-missing baseline and at least 1 post-baseline BRIEF-A:Self Report result within each group, Last Observation Carried Forward (LOCF) were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 187 | 173
units on a scale | -5.70 (1.88) | 0.90 (1.81)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.006, ANCOVA

7. Secondary Outcome: Change From Baseline in the Behavior Rating Inventory of Executive Function-Adult Version:Informant Report (BRIEF-A:Informant) Global Executive Composite (GEC) Index Score From Week 24 to Week 49
Description: BRIEF-A:Informant is a 75-item third-party observer's view of the participants' executive functions/self-regulation in their everyday environment. Items include: Inhibit, Shift, Emotional Control, Self Monitor, Initiate, Working Memory, Plan/Organize, Task Monitor, and Organization of Materials. Behavior is rated on a 3-point scale: 1 (behavior is never observed) to 3 (behavior is often observed). GEC Index Score is a subscore of the 75-item BRIEF-A score, reflects overall functioning and was calculated based on 70 items. Total scores range: 70-210. Lower scores = less perceived impairment. Least Squares (LS) Mean values were adjusted for treatment, pooled Investigator, and baseline.
Time Frame: Baseline (Week 24), Week 49
Population: Participants with a non-missing baseline and at least 1 post-baseline BRIEF-A:Informant result within each group, Last Observation Carried Forward (LOCF) were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 154 | 147
units on a scale | -8.4 (2.16) | -0.6 (2.17)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.006, ANCOVA

8. Secondary Outcome: Change From Baseline in European Quality of Life (EuroQoL) Questionnaire-5 Dimensions (EQ-5D) Index Score From Week 24 to Week 49
Description: The EQ-5D is a Self-reported, 5-item scale to assess health utility (mobility, self-care, usual activities, pain and discomfort, and depression/anxiety). Scoring is on a 3-point scale (1=no health problems, 2=some or moderate problems, 3=major health problems). A preference value Index score is calculated using societal preference developed from a general population-based valuation studies. Index score ranges: United Kingdom (UK): -0.59 to 1.0, United States (US): -0.11 to 1.0, where 1 represents best possible health and 0 represents dead, with <0 interpreted as a health state "worse than dead." A Quality of Life Health State Score visual analog scale (VAS) was assessed, scores range from 0 to 100. Higher scores indicate better health state. Least Square (LS) Mean values were adjusted for treatment, pooled Investigator, baseline.
Time Frame: Baseline (Week 24), Week 49
Population: Participants with a non-missing baseline and at least 1 post-baseline EQ-5D Index Score or VAS score within each group, Last Observation Carried Forward (LOCF) were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 197 | 180
units on a scale
  UK population-based Index Score (n=194, 180) | 0.00 (0.01) | 0.00 (0.01)
  US population-based Index Score (n=194, 180) | 0.00 (0.01) | 0.00 (0.01)
  Health State Score (N=197, 179) | 4.60 (1.21) | 3.20 (1.19)

ADVERSE EVENTS:
Groups:
- Atomoxetine (Study Periods 2 and 3A): 40-100 milligrams/day (mg/day) atomoxetine orally, once daily or twice daily for 12 weeks during open-label, acute-treatment phase (Study Period 2), and 80-100 mg/day for 12 weeks during double-blind maintenance phase of Study Period 3 (Study Period 3A).
- Atomoxetine (Study Period 3B): 40-100 milligrams/day (mg/day) atomoxetine orally, once daily or twice daily for 12 weeks during open-label, acute-treatment phase (Study Period 2), and 80-100 mg/day for 12 weeks during double-blind maintenance phase of Study Period 3 (Study Period 3A).
  Followed by 80-100 mg/day atomoxetine orally, once daily or twice daily for 25 weeks during double-blind randomized withdrawal phase of Study Period 3 (Study Period 3B).
- Placebo (Study Period 3B): 40-100 milligrams/day (mg/day) atomoxetine orally, once daily or twice daily for 12 weeks during open-label, acute-treatment phase (Study Period 2), and 80-100 mg/day for 12 weeks during double-blind maintenance phase of Study Period 3 (Study Period 3A).
  Followed by Placebo orally, once daily or twice daily for 25 weeks during double-blind randomized withdrawal phase of Study Period 3 (Study Period 3B).
- Atomoxetine (Study Period 4; Open-Label Extension): 40-100 milligrams/day (mg/day) atomoxetine orally, once daily or twice daily for 12 weeks during open-label, acute-treatment phase (Study Period 2), and 80-100 mg/day for 12 weeks during double-blind maintenance phase of Study Period 3 (Study Period 3A) and for 25 weeks during double-blind randomized withdrawal phase of Study Period 3 (Study Period 3B), followed by a 2 year open label extension (Study Period 4). The open-label extension was optional and only offered to participants living in countries where atomoxetine for the adult ADHD indication had not been approved who had completed the Study Period 3B and were receiving benefit from the drug.
Arm/Group | Atomoxetine (Study Periods 2 and 3A) | Atomoxetine (Study Period 3B) | Placebo (Study Period 3B) | Atomoxetine (Study Period 4; Open-Label Extension)
Serious Adverse Events (participants affected / at risk) | 29/2011 | 7/266 | 3/258 | 14/180
Other Adverse Events (participants affected / at risk) | 1611/2011 | 120/266 | 96/258 | 119/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine (Study Periods 2 and 3A) (N=2011) | Atomoxetine (Study Period 3B) (N=266) | Placebo (Study Period 3B) (N=258) | Atomoxetine (Study Period 4; Open-Label Extension) (N=180)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hepatitis alcoholic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Diaphragmatic injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Splenic injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressive symptom (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hallucination, auditory (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bunion operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin neoplasm excision (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine (Study Periods 2 and 3A) (N=2011) | Atomoxetine (Study Period 3B) (N=266) | Placebo (Study Period 3B) (N=258) | Atomoxetine (Study Period 4; Open-Label Extension) (N=180)
Angina pectoris (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0) | 3 (3)
Palpitations (Cardiac disorders) | 83 (90) | 1 (1) | 1 (1) | 2 (2)
Tachycardia (Cardiac disorders) | 70 (73) | 3 (4) | 1 (1) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 38 (46) | 0 (0) | 1 (1) | 3 (4)
Conjunctivitis (Eye disorders) | 8 (8) | 0 (0) | 1 (1) | 2 (2)
Vision blurred (Eye disorders) | 32 (32) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 29 (30) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 38 (41) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 61 (73) | 2 (2) | 2 (2) | 3 (3)
Constipation (Gastrointestinal disorders) | 93 (99) | 1 (1) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 53 (60) | 4 (4) | 5 (5) | 8 (10)
Dry mouth (Gastrointestinal disorders) | 342 (368) | 3 (4) | 2 (2) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 65 (72) | 1 (1) | 0 (0) | 6 (6)
Gastritis (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0) | 6 (6)
Haemorrhoids (Gastrointestinal disorders) | 4 (5) | 1 (1) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 552 (707) | 6 (6) | 3 (4) | 9 (9)
Toothache (Gastrointestinal disorders) | 23 (25) | 1 (1) | 2 (2) | 1 (2)
Vomiting (Gastrointestinal disorders) | 82 (96) | 1 (1) | 3 (3) | 1 (1)
Chills (General disorders) | 57 (60) | 0 (0) | 0 (0) | 2 (2)
Fatigue (General disorders) | 262 (292) | 1 (1) | 3 (3) | 4 (5)
Influenza like illness (General disorders) | 11 (11) | 2 (3) | 1 (1) | 2 (2)
Irritability (General disorders) | 80 (87) | 2 (2) | 0 (0) | 0 (0)
Malaise (General disorders) | 46 (57) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 16 (17) | 4 (4) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 18 (19) | 3 (3) | 2 (2) | 5 (7)
Cystitis (Infections and infestations) | 8 (8) | 1 (1) | 1 (1) | 5 (8)
Ear infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 24 (24) | 5 (5) | 2 (2) | 5 (7)
Gastrointestinal infection (Infections and infestations) | 4 (4) | 0 (0) | 0 (0) | 2 (2)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 52 (55) | 8 (8) | 6 (6) | 10 (10)
Nasopharyngitis (Infections and infestations) | 137 (153) | 18 (26) | 13 (16) | 22 (39)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Rhinitis (Infections and infestations) | 13 (13) | 1 (1) | 2 (2) | 4 (4)
Sinusitis (Infections and infestations) | 23 (24) | 2 (2) | 3 (4) | 4 (4)
Tonsillitis (Infections and infestations) | 9 (9) | 1 (1) | 2 (2) | 3 (4)
Upper respiratory tract infection (Infections and infestations) | 57 (62) | 11 (13) | 7 (7) | 1 (2)
Urinary tract infection (Infections and infestations) | 12 (12) | 1 (2) | 0 (0) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 8 (8) | 5 (5) | 0 (0) | 0 (0)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 1 (1) | 2 (2)
Blood pressure increased (Investigations) | 13 (13) | 4 (6) | 0 (0) | 3 (3)
Heart rate increased (Investigations) | 21 (24) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 39 (39) | 1 (1) | 1 (1) | 2 (2)
Weight increased (Investigations) | 13 (13) | 3 (3) | 1 (1) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 294 (319) | 1 (1) | 1 (1) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 10 (10) | 1 (1) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 (15) | 2 (2) | 1 (1) | 8 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 30 (30) | 3 (3) | 7 (7) | 7 (9)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1) | 1 (1) | 2 (2)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 170 (195) | 1 (1) | 2 (2) | 3 (3)
Headache (Nervous system disorders) | 347 (482) | 13 (15) | 11 (11) | 17 (38)
Migraine (Nervous system disorders) | 26 (46) | 1 (3) | 1 (1) | 3 (3)
Paraesthesia (Nervous system disorders) | 74 (76) | 1 (1) | 0 (0) | 2 (2)
Sedation (Nervous system disorders) | 26 (27) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 112 (126) | 1 (1) | 1 (1) | 1 (2)
Tremor (Nervous system disorders) | 25 (26) | 0 (0) | 1 (1) | 3 (3)
Abnormal dreams (Psychiatric disorders) | 34 (35) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 28 (32) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 60 (62) | 3 (3) | 3 (3) | 2 (2)
Depressed mood (Psychiatric disorders) | 56 (62) | 0 (0) | 2 (2) | 4 (5)
Depression (Psychiatric disorders) | 34 (34) | 2 (2) | 3 (4) | 1 (1)
Initial insomnia (Psychiatric disorders) | 34 (40) | 4 (4) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 177 (209) | 3 (3) | 1 (1) | 4 (6)
Libido decreased (Psychiatric disorders) | 61 (65) | 2 (2) | 2 (2) | 1 (1)
Middle insomnia (Psychiatric disorders) | 33 (35) | 2 (2) | 0 (0) | 3 (3)
Nervousness (Psychiatric disorders) | 9 (9) | 1 (1) | 0 (0) | 2 (3)
Restlessness (Psychiatric disorders) | 27 (34) | 1 (1) | 0 (0) | 2 (3)
Sleep disorder (Psychiatric disorders) | 71 (82) | 1 (1) | 1 (1) | 5 (5)
Dysuria (Renal and urinary disorders) | 49 (54) | 1 (1) | 0 (0) | 2 (2)
Urinary hesitation (Renal and urinary disorders) | 43 (46) | 2 (2) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 21 (22) | 0 (0) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 19 (23) | 1 (2) | 1 (1) | 2 (2)
Ejaculation disorder (Reproductive system and breast disorders) | 25 (29) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 99 (103) | 3 (3) | 0 (0) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 22 (23) | 5 (6) | 1 (1) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 20 (20) | 5 (5) | 4 (5) | 6 (6)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 1 (1) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 180 (196) | 2 (2) | 0 (0) | 8 (8)
Piloerection (Skin and subcutaneous tissue disorders) | 23 (25) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 12 (12) | 1 (1) | 0 (0) | 2 (2)
Tooth extraction (Surgical and medical procedures) | 5 (7) | 0 (0) | 1 (1) | 2 (2)
Hot flush (Vascular disorders) | 56 (61) | 3 (3) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 27 (28) | 1 (1) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days